CLINICAL TRIAL: NCT01988116
Title: Vitamin D Replacement in Chronic Kidney Disease and Its Effects on Iron Homeostasis, Serum Hepcidin, and Hemojuvelin Levels.
Brief Title: Effects of Vitamin D Replacement on Hormones Regulating Iron Metabolism in Individuals With Chronic Kidney Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: F130725013
Record Dates: First submitted 2013-11-04; First posted 2013-11-20 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Kidney Disease; Anemia of Chronic Disease
Keywords: Chronic kidney disease; Anemia of chronic disease; Iron Metabolism; Iron Homeostasis; Vitamin D; Calcitriol; hemojuvelin; hepcidin; anemia; ferroportin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Calcitriol (Experimental): Oral Calcitriol 0.5 mcg once daily for 6 weeks
  Interventions: Drug: Oral Calcitriol 0.5 mcg once daily for 6 weeks
- Placebo Arm (Placebo Comparator): Placebo capsule 1 Capsule once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Calcitriol 0.5 mcg once daily for 6 weeks
  Other Names: Rocaltrol
  Arms: Oral Calcitriol
Drug: Placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of the study is to learn more about how treatment with vitamin D can affect iron metabolism and blood levels of two hormones that control iron levels, hepcidin and hemojuvelin in people with chronic kidney disease (CKD).

Iron is an essential mineral which is a major component of proteins that carry oxygen in the blood. Problems with iron metabolism can lead to low blood levels (anemia), which can commonly happen in people with CKD.

New research over the last decade has uncovered a new hormone called 'hepcidin', which is made in the liver and released into the blood. Hepcidin controls how much iron is in the blood by preventing the absorption of iron from food. Blood levels of hepcidin C are found to be high in people with CKD, and a recent small study in people with normal kidney function showed that treatment with vitamin D decreased hepcidin levels.

Another protein, known as 'hemojuvelin', has been recently discovered and is also thought to control the amount of iron in the blood. The relationship between vitamin D and hemojuvelin has never been studied before.

In this study, investigators would like to examine the effects of vitamin D on iron metabolism and blood levels of hepcidin C and hemojuvelin in individuals with CKD.

DETAILED DESCRIPTION:
Iron homeostasis is tightly regulated in humans. Iron is mostly recycled from hemoglobin, myoglobin and other enzymes. Since humans lack the capacity to excrete excess iron, it must be intricately regulated at the site of its absorption in the duodenum and proximal jejunum. In the last decade, hepcidin has emerged as a master regulator of iron homeostasis. It decreases iron absorption from the gut mucosa by limiting its transport from the enterocyte across the basolateral membrane into the circulation. It does so by down-regulating the synthesis or promoting internalization of a basolateral membrane protein 'Ferroportin', the only known cellular iron exporter.

Vitamin D is hypothesized to exert a significant and independent effect on the iron metabolism. In the CKD population, low vitamin-D levels independently correlate with the severity of anemia. Hepcidin C levels are found to be elevated in the CKD population. Mechanisms underlying the effect of vitamin D on iron homeostasis potentially include vitamin D induced expression of erythropoietin receptors, increased proliferation of erythroid precursors, and reduction in hepcidin C levels due to reduction in IL-6 from the anti-inflammatory effects of vitamin D. More recently, a study revealed direct relationship between vitamin D replacement and a sustained fall in hepcidin C levels. The same group of researchers found the above relationship to be due to a direct effect of vitamin D on hepcidin expression.

Hemojuvelin (HJV) is a protein encoded by the HFE2 gene and is found in the membrane bound and the soluble form (sHJV) in the humans. Mutations in the HJV gene are responsible for Juvenile Hemochromatosis. It is an upstream regulator of hepcidin transcription and appears to be essential for hepcidin expression in the hepatocytes and has important role to play in iron homeostasis. Recently, an assay has become available to measure the sHJV levels in the serum.

Although, we know that hepcidin plays a central role in iron homeostasis and recent studies have given us insight into the role hemojuvelin and vitamin D play in iron metabolism, to date, no studies have examined the effect on vitamin D replacement on hepcidin, hemojuvelin levels and iron metabolism in individuals with CKD.

Hypothesis 1: Treatment with an activated vitamin D analog in the individuals with CKD results in a statistically significant fall in hepcidin C levels as compared to individuals provided with placebo.

Hypothesis 2: Treatment with an activated vitamin D analog results in decreased levels of soluble hemojuvelin in individuals with chronic kidney disease.

Hypothesis 3: Vitamin D replacement in the individuals with CKD results in improved iron parameters as compared to the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate CKD (eGFR 15 - 60 ml/min/1.73 m2) as estimated by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula.

Exclusion Criteria:

* Subjects currently receiving active vitamin D analog therapy or history of recent (< 3 months) use.
* Subjects currently receiving nutritional vitamin D (cholecalciferol or ergocalciferol) in dosages greater than 2000 IU/day.
* Subjects receiving erythropoiesis stimulating agents.
* Subjects receiving intravenous iron therapy.
* Subjects receiving oral iron therapy started within 3 months prior to recruitment.
* Subjects with severe anemia defined as Hb < 8.0 g/dL for males and Hb <7.0 g/dL for females.
* Subjects with iron deficiency anemia defined as serum ferritin <100ng/ml and Transferring Saturation < 20%.
* Pregnancy and lactation.
* Subjects with hypercalcemia defined as serum calcium level of > 10.0 mg/dL.
* Subjects with serum phosphorus concentration of > 4.5 mg/dL.
* Subjects with acute kidney injury or rapidly declining GFR.
* Subjects receiving any form of renal replacement therapy including hemodialysis, peritoneal dialysis, and patients with renal transplant.
* Subjects with focus of active inflammation or infection determined clinically.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in serum hepcidin levels | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
Change in soluble hemojuvelin | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
Change in other indices of iron metabolism | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
  Including, Serum Ferritin, Iron level, Percent transferrin saturation and TIBC

SECONDARY OUTCOMES:
Change in serum hemoglobin | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bhupesh Panwar, MD, Principal Investigator — University of Alabama, Nephrology Division; Orlando M Gutierrez, MD,MMSc, Study Director — University of Alabama, Nephrology Division
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Panwar B, McCann D, Olbina G, Westerman M, Gutierrez OM. Effect of calcitriol on serum hepcidin in individuals with chronic kidney disease: a randomized controlled trial. BMC Nephrol. 2018 Feb 9;19(1):35. doi: 10.1186/s12882-018-0823-7. PMID 29426300